CLINICAL TRIAL: NCT06412185
Title: A Randomized, Double-blind, Placebo-controlled Phase I Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Single Dose Escalation of CM383 in Male Healthy Subjects
Brief Title: Single Dose Escalation Study of CM383 in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM383-100001
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (Experimental): CM383 injection and matched placebo, intravenous injection
  Interventions: Biological: CM383; Other: Placebo
- Group 2 (Experimental): CM383 injection and matched placebo, intravenous injection
  Interventions: Biological: CM383; Other: Placebo
- Group 3 (Experimental): CM383 injection and matched placebo, intravenous injection
  Interventions: Biological: CM383; Other: Placebo
- Group 4 (Experimental): CM383 injection and matched placebo, intravenous injection
  Interventions: Biological: CM383; Other: Placebo
- Group 5 (Experimental): CM383 injection and matched placebo, intravenous injection
  Interventions: Biological: CM383; Other: Placebo
- Group 6 (Experimental): CM383 injection and matched placebo, intravenous injection
  Interventions: Biological: CM383; Other: Placebo

INTERVENTIONS:
Biological: CM383 — CM383 Injection
Other: Placebo — Placebo

SUMMARY:
This study is a single center, randomized, double-blind, placebo-controlled Phase I clinical study in a single dose escalation to evaluate its safety, tolerability, pharmacokinetics, pharmacodynamics, and immunogenicity of CM383 in male healthy subjects.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is the most common type of dementia, which is a degenerative disease of the central nervous system with insidious onset and progressive development. Its clinical features mainly include memory impairment, cognitive impairment, psychobehavioral abnormalities, and social decline.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males, voluntarily participate;
* 18 and 80 years old (including boundary values);
* able to communicate well with the researchers and follow up the protocol requirements.

Exclusion Criteria:

* The average daily smoking volume within three months before screening is greater than 5 cigarettes;
* Excessive alcohol consumption within three months before screening, or positive alcohol breath test;
* Urine drug abuse screening is positive;
* Having a family planning or sperm donation plan; Disagree to adopt efficient contraceptive measures.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Up to week 12
  Incidence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Wen, Principal Investigator — Jinan Central Hospital
Locations (1):
- Jinan Central Hospital, Jinan, Shandong, China